CLINICAL TRIAL: NCT05732025
Title: Evaluation of Safety and Effectiveness of the SONICO-CX Intracoronary Electrohydraulic Shockwave Balloon Catheter/Hydraulic Shock Wave Lithotripsy, A Prospective, Single-center, Randomized Controlled Exploratory Clinical Study
Brief Title: Evaluation of Safety and Effectiveness of the SONICO-CX Intracoronary Electrohydraulic Shockwave Balloon Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT020
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-07

CONDITIONS: Calcified Atheroma
Keywords: Calcified coronary lesions; Rotary atherectomy; Electrohydraulic shock wave lithotripsy; Optical coherence tomography (OCT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrohydraulic shock wave lithotripsy (Experimental): Pre-treatment of severe calcified coronary lesions with electrohydraulic shock wave lithotripsy
  Interventions: Device: Electrohydraulic shock wave lithotripsy
- Rotary atherectomy (Active Comparator): Pre-treatment of severe calcified coronary lesions with Rotary atherectomy
  Interventions: Device: Rotary atherectomy

INTERVENTIONS:
Device: Electrohydraulic shock wave lithotripsy — Pre-treatment of severe calcified coronary lesions with electrohydraulic shock wave lithotripsy
  Arms: Electrohydraulic shock wave lithotripsy
Device: Rotary atherectomy — Pre-treatment of severe calcified coronary lesions with rotary atherectomy
  Arms: Rotary atherectomy

SUMMARY:
Calcified coronary lesions often run through various complex lesions, which increases the difficulty of coronary intervention, is one of the main challenges faced by interventional cardiovascular physicians. Severely calcified lesions, or severely calcified lesions with twisted, angulated, diffused, significantly increase rates of immediate complications and early and late major adverse cardiovascular events. Correctly identifying and evaluating calcified lesions, and selecting the most appropriate treatment strategy according to the degree of coronary artery calcification are very important for improving the success rate of intervention, reducing complications, and improving the short-term and long-term prognosis of patients.

DETAILED DESCRIPTION:
Calcified coronary lesions often run through various complex lesions, which increases the difficulty of coronary intervention, is one of the main challenges faced by interventional cardiovascular physicians. Severely calcified lesions, or severely calcified lesions with twisted, angulated, diffused, significantly increase rates of immediate complications and early and late major adverse cardiovascular events. Correctly identifying and evaluating calcified lesions, and selecting the most appropriate treatment strategy according to the degree of coronary artery calcification are very important for improving the success rate of intervention, reducing complications, and improving the short-term and long-term prognosis of patients.The current regular interventional treatment methods for coronary calcification lesions include plain balloons, non-compliant balloons, cutting balloons, etc., but the incidence of complications is high and the rate of long-term restenosis is high, and the effect is not satisfactory. Rotary atherectomy is currently the main pretreatment method for severe calcified lesions. Rotary atherectomy combined with drug-eluting stent implantation has become an important mean for the treatment of severe calcified lesions, even complex lesions, in the DES era, and has good safety and effectiveness. However, this technique is more complicated, and in order to ensure its advantages, it needs correct and meticulous operation by an experienced interventional team. Studies have shown that the use rate of rotational atherectomy in high-capacity centers is only 3% to 5%. The reasons may be related to the expensive equipment, difficult operation and unfamiliarity with new technologies. The intra-coronary electrohydraulic shock wave balloon catheter is a device that combines electrohydraulic shock wave lithotripsy with percutaneous transluminal angioplasty. After the catheter is connected to the device and energized, the micro-transmitter installed in the balloon can generate pulsed sound pressure waves to shatter the calcified plaque inside the target lesion, enabling subsequent expansion of the lesion at low pressure. SONICO-CX intracoronary electrohydraulic shock wave balloon catheter is a new type of plaque remodeling device, which can not only change the compliance of the artery, but also reduce the damage of the vessel wall. It provides a new option for doctors to better solve the problem of severe calcified lesions, and also brings more benefits to patients. This randomized trial was conducted to assess the efficacy/safety of intracoronary electrohydraulic shock wave lithotripsy versus rotational atherectomy based on optical coherence tomography (OCT) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria:

  1. Age ≥ 18 years old
  2. Evidence of asymptomatic ischemia, stable or unstable angina
  3. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent, and are willing to accept angiography, OCT examination and clinical follow-up.
* Angiographic Criteria:

  1. The target lesion is primary and in situ coronary artery lesion
  2. The length of the target lesion is ≤60mm, and the diameter of the target lesion is 2.5-4.0mm (visually)
  3. The stenosis rate of the target lesion diameter is ≥70%, and the doctor judges that it is necessary to implant a stent (visual inspection method) to meet one of the following:

     1. Diameter stenosis ≥ 70%, < 100%
     2. ≥50%, <70% with evidence of ischemia
  4. The lesion allows a 0.014 guidewire to pass
  5. Under multi-angle imaging conditions, calcified shadow lesions can be seen on both sides of the lesion vessel wall (the target lesion meets the definition of severe calcification)

Exclusion Criteria:

* Clinical Criteria:

  1. Acute myocardial infarction occurred within 30 days before operation
  2. Use special balloons (chocolate balloons, scored balloons, spinous balloons, etc.) to treat lesions at the same time
  3. Troponin is greater than 5 times the upper limit of laboratory normal value within one week before operation
  4. Severe cardiac dysfunction (grade III or IV)
  5. Left ventricular ejection fraction <25%
  6. The patient refuses emergency CABG surgery or does not have indications for emergency CABG surgery
  7. Severe uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg)
  8. Severe renal failure (serum creatinine > 221 μmol/L)
  9. Preoperative hemoglobin <100g/L
  10. Obvious coagulation dysfunction (platelet count<100×109/L or INR>1.7, INR is only required for patients who have taken warfarin orally within 2 weeks before enrollment)
  11. Blood hypercoagulability diseases (such as polycythemia vera, platelet count >750×109/L, etc.)
  12. History of stroke or TIA within 3 months
  13. History of active peptic ulcer or upper gastrointestinal bleeding within 6 months
  14. The life expectancy of the patient is less than 12 months
  15. The patient has an active systemic infection
  16. The patient has a connective tissue disorder (such as Marfan syndrome)
  17. Patient is allergic to contrast material
  18. Patients undergoing heart transplantation
  19. Patients with implanted cardiac pacemakers
  20. The patient is pregnant or breastfeeding
  21. Those who have participated in clinical trials of other drugs or medical devices within one month before enrollment;
  22. Other circumstances that the investigator considers inappropriate to participate in the trial
* Angiographic Criteria:

  1. Unprotected left main lesion (left main visual stenosis >50%)
  2. Baseline TIMI blood flow is less than grade 3 (evaluation after pre-dilation is allowed)
  3. A stent has been implanted within 10mm of the proximal or distal end of the target lesion
  4. The target lesion is located distal to the saphenous vein or LIMA/RIMA bypass graft
  5. Aneurysm in the target vessel
  6. Angiography confirmed the presence of thrombus in the target vessel
  7. Chronic total occlusive disease
  8. Angiography confirmed the presence of severe dissection of the target lesion before hydroelectric shock wave lithotripsy (D-F type dissection (NHLBI classification)
  9. The investigator judged that the target lesion is not suitable for patients with vasodilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Stent expansion rate using OCT | Immediately after surgery
  Stent expansion rate=Minimum lumen area in the stent/(distal reference vessel area + proximal reference vessel area)*1/2

SECONDARY OUTCOMES:
Angiography success rate | Immediately after surgery
Minimum stent area (MSA) immediately after surgery | Immediately after surgery
Minimum lumen diameter MLD immediately after operation | Immediately after surgery
The diameter of the lumen immediately after operation | Immediately after surgery
Obtained lumen area immediately after operation | Immediately after surgery
Lumen acquisition rate immediately after operation | Immediately after surgery
Incomplete apposition rate of stent | Immediately after surgery
Symmetry of the expansion of stent | Immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Zhejiang University, School of Medicine

IPD SHARING:
Plan to Share IPD: No